CLINICAL TRIAL: NCT03156478
Title: STOP DIABETES - Knowledge-based Solutions
Acronym: StopDia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: National Institute of Health and Welfare (Unknown); Technical Research Centre of Finland (Unknown); University of Melbourne (Other); University of Konstanz (Other); Karolinska Institutet (Other); Maastricht University (Other); University of Oslo (Other); Danube-University (Unknown); Flinders University (Other); Cornell University (Other); University of Copenhagen (Other); Roskilde University (Other); University of Manchester (Other); University of York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 467/2016
Record Dates: First submitted 2017-04-13; First posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Type2 Diabetes; Life Style; Diet Habit; Physical Activity; Empowerment
Keywords: Prevention; Digital solutions; Type 2 diabetes; Life style modification; Physical activity; Healthy diet; Health economics; Environmental choice architecture; Socio-economic facilitators; Socio-economic barriers; Wellbeing
MeSH Terms: conditions — Feeding Behavior; Motor Activity; Empowerment; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Participants will be randomized in 3 groups: 1) control group, 2) digital lifestyle intervention group and 3) combined digital and face-to-face lifestyle intervention group. Environmental changes will be done within some work places.Part of the participants in each group may be exposed to environmental modification that are aimed for lifestyle changes at work places.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): At baseline, individuals in the control group receive digital information package about lifestyle risk factors of type 2 diabetes with recommendations on healthy diet and physical activity in accordance with the Finnish Nutrition Recommendations and the national recommendation for health enhancing physical activity.
- Digital lifestyle intervention group (Experimental): Participants are instructed to use a digital self-help tool for 12 months. This tool is developed in the StopDia-study to enact positive changes in participant's health behaviour. The digital intervention consists of 2 components which motivate, enable and trigger the participants to improve their health behaviours. B.J. Fogg's Tiny Habits -ideology. The digital intervention is based on the Fogg Behaviour Model (FBM) and the Behaviour Wizard.
  Interventions: Behavioral: Digital lifestyle intervention group
- Combined digital and face-to-face lifestyle intervention group (Experimental): Participants are using the StopDia digital solution tool as described above. In addition, they have six face-to-face group coaching (6-15 participants/group) sessions at local health centers facilitated by trained nurses. The face-to-face group intervention is based on the Self-Determination Theory and theories of self-regulation, and delivered using intrinsic motivational coaching approach designed and tested in the GOAL lifestyle intervention, and further developed in several other studies in Finland and internationally.
  Interventions: Behavioral: Combined digital and face-to-face lifestyle intervention group

INTERVENTIONS:
Behavioral: Digital lifestyle intervention group — Intervention with digital application for lifestyle changes
  Arms: Digital lifestyle intervention group
Behavioral: Combined digital and face-to-face lifestyle intervention group — Intervention with digital application and group meetings for lifestyle changes
  Arms: Combined digital and face-to-face lifestyle intervention group

SUMMARY:
The aim of the Stop Diabetes - Knowledge based solutions (StopDia) consortium project (University of Eastern Finland, National Institute for Health and Welfare, and Technical Research Centre of Finland) is to develop and test approaches to identify individuals at increased risk of type 2 diabetes and to empower them in adopting and maintaining a healthy lifestyle by combining individual and environment level strategies into a dual-process approach targeting deliberative and automatic processes of behavior. We also aim to identify barriers and facilitators of adopting a healthy lifestyle in the society, create a model for the prevention of type 2 diabetes by joint actions of health care, third sector, and other societal actors, and develop methods to monitor the cost-effectiveness of these actions. We will carry out a 1-year randomized controlled trial on the effects of among 10 000 individuals aged 18-70 years at increased risk of type 2 diabetes living in Finland. The participants will be randomized into the control group, the digital lifestyle intervention group, or the combined digital and face-to-face lifestyle intervention group. The aim of the interventions is to enhance diet quality, increase physical activity, decrease body weight, and improve glucose tolerance in individuals at increased risk of type 2 diabetes.

DETAILED DESCRIPTION:
Type 2 diabetes is a major public health and economical problem all over the world, including Finland. A healthy diet and physical activity are the cornerstones for the prevention of type 2 diabetes. The aim of the Stop Diabetes - Knowledge based solutions (StopDia) study is to develop and test approaches to identify individuals at increased risk of type 2 diabetes and to empower them in adopting and maintaining a healthy lifestyle by combining individual and environment level strategies into a dual-process approach targeting deliberative and automatic processes of behavior. We also aim to identify barriers and facilitators of adopting a healthy lifestyle in the society, create a model for the prevention of type 2 diabetes by joint actions of health care, third sector, and other societal actors, and develop methods to monitor the cost-effectiveness of these actions. We will recruit 10 000 individuals aged 18-70 years at increased risk of type 2 diabetes living in the hospital district of Northern Savo, Päijät-Häme, or South Karelia in Finland for a 1-year randomized controlled trial. We will assess body height and weight, body mass index, waist circumference, and blood pressure, take blood samples for biochemical analyses, and perform a 2-hour oral glucose tolerance test at baseline. The participants will be asked to fill out a detailed digital questionnaire on factors related to the risk of type 2 diabetes, including diet, physical activity, sedentary behavior, health status, physical, psychic, and social well-being, as well as the use of health care services and medications. The participants will be randomized into the control group, the digital lifestyle intervention group, or the combined digital and face-to-face lifestyle intervention group. The aim of the interventions is to enhance diet quality, increase physical activity, decrease body weight, and improve glucose tolerance in individuals at increased risk of type 2 diabetes. We will also investigate the effects of environmental interventions at certain workplaces and the synergistic effects of the individual level and environmental interventions in a subsample of the study population. All baseline assessments will be repeated after the 1-year follow-up. The primary outcomes will be the changes in diet, total physical activity, body weight, and plasma glucose levels from the oral glucose tolerance test. After the 1-year intervention study, follow-up examinations will be performed 3, 5, 10, 15, and 20 years after the baseline examinations.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-70 years
* 12 points or more in the Finnish diabetes risk score or previous gestational diabetes or repeated impaired fasting glucose (IFG) (fasting plasma glucose level 6,1 - 6,9 mmol/l) or impaired glucose tolerance (2-hour glucose level 7,8 - 11,0 mmol/l in oral glucose tolerance test)
* living in the hospital district of Northern Savo, Päijät-Häme or South Karelia
* possibility to use computer, smartphone or tablet with internet connection
* having own self-phone number
* adequate Finnish language skill

Exclusion Criteria:

* type 1 or 2 diabetes
* pregnancy or breastfeeding
* current cancer or less than 6 months from the end of cancer treatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Change in diet | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Change in diet is assessed by the dietary score based on Finnish Nutrition Recommendations and is formulated according to food frequency questionnaire.
Change in total physical activity level | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Change in total physical activity level is assessed by the physical activity questionnaire.
Change in plasma glucose levels | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed in the 2 hour oral glucose tolerance tests
Change in body weight | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed with digital weight scales

SECONDARY OUTCOMES:
Change in waist circumference | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed with validated guidelines for the measure
Change in insulin concentration | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed in the 2 hour oral glucose tolerance tests
Change in glycated hemoglobin | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed from fasting blood sample
Change in plasma lipid concentration | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Plasma total, HDL and LDL cholesterol, and triglyceride concentrations are measured.
Change in resting blood pressure | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up.
  Resting systolic and diastolic blood pressure is measured by automatic sphygmomanometer in sitting position.
Change in inflammation markers | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up.
  Serum high-sensitivity C-reactive protein (hs-CRP) and interleukine-1Ra (IL-1Ra) are measured as biomarkers of inflammation.
Change in liver function | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up.
  Plasma aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are measured as biomarkers of liver function.
Change in metabolite profiles | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Metabolites and metabolic profiles related to diet, other lifestyle factors and predicting type 2 diabetes measured from serum and plasma samples
Change in sedentary behavior | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Change in sedentary behavior is described as the total amount spent in sitting and lying position during waking hours, and is assessed by the questionnaire.
Change in sleeping behavior | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Formulated according to sleeping behavior questionnaire
Change in smoking behavior | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed by questionnaire
Change in alcohol consumption | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Assessed by food frequency questionnaire
Change in eating behavior | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Eating behavior is assessed by questionnaires.
Change in mental wellbeing | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Change in mental wellbeing is assessed by questionnaire.
Change in quality of life | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up.
  Quality of life is assessed by questionnaire.
Use of health-care services and associated costs | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up
  Use of health-care services are assessed by questionnaire and registers. Associated costs are calculated based on these data.
Work ability and associated costs | From baseline to one year follow-up, to 3 year follow-up, to 5 year follow-up, to 10 year follow-up, to 15 year follow-up, 20 year follow-up.
  Work ability is assessed by questionnaire. Associated costs are calculated based on these data.
User experience of the Internet intervention | During the intervention at the time point of two weeks, and at one year follow-up
  Measured by the questionnaires.
Usage of the Internet intervention | During the intervention at the time point of two weeks, 3 months, 6 months, and at one year follow-up
  Measured by the log data

CONTACTS AND LOCATIONS:
Overall Officials: Jussi Pihlajamäki, MD, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lakka TA, Aittola K, Jarvela-Reijonen E, Tilles-Tirkkonen T, Mannikko R, Lintu N, Karhunen L, Kolehmainen M, Harjumaa M, Mattila E, Jarvenpaa R, Ermes M, Mikkonen S, Martikainen J, Poutanen K, Schwab U, Absetz P, Lindstrom J, Pihlajamaki J. Real-world effectiveness of digital and group-based lifestyle interventions as compared with usual care to reduce type 2 diabetes risk - A stop diabetes pragmatic randomised trial. Lancet Reg Health Eur. 2023 Jan;24:100527. doi: 10.1016/j.lanepe.2022.100527. Epub 2022 Oct 12. PMID 36620354
- [Derived] Lavikainen P, Mattila E, Absetz P, Harjumaa M, Lindstrom J, Jarvela-Reijonen E, Aittola K, Mannikko R, Tilles-Tirkkonen T, Lintu N, Lakka T, van Gils M, Pihlajamaki J, Martikainen J. Digitally Supported Lifestyle Intervention to Prevent Type 2 Diabetes Through Healthy Habits: Secondary Analysis of Long-Term User Engagement Trajectories in a Randomized Controlled Trial. J Med Internet Res. 2022 Feb 24;24(2):e31530. doi: 10.2196/31530. PMID 35200147
- [Derived] Karlund A, Kaariainen T, Kostamo VM, Kokkola T, Kolehmainen M, Lakka TA, Pihlajamaki J, Manninen A. Oxygen-18 and carbon-13 isotopes in eCO2and erythrocytes carbonic anhydrase activity of Finnish prediabetic population. J Breath Res. 2021 Jan 22;15(2). doi: 10.1088/1752-7163/abd28d. PMID 33302264
- [Derived] Harjumaa M, Absetz P, Ermes M, Mattila E, Mannikko R, Tilles-Tirkkonen T, Lintu N, Schwab U, Umer A, Leppanen J, Pihlajamaki J. Internet-Based Lifestyle Intervention to Prevent Type 2 Diabetes Through Healthy Habits: Design and 6-Month Usage Results of Randomized Controlled Trial. JMIR Diabetes. 2020 Aug 11;5(3):e15219. doi: 10.2196/15219. PMID 32779571
- [Derived] Pihlajamaki J, Mannikko R, Tilles-Tirkkonen T, Karhunen L, Kolehmainen M, Schwab U, Lintu N, Paananen J, Jarvenpaa R, Harjumaa M, Martikainen J, Kohl J, Poutanen K, Ermes M, Absetz P, Lindstrom J, Lakka TA; StopDia study group. Digitally supported program for type 2 diabetes risk identification and risk reduction in real-world setting: protocol for the StopDia model and randomized controlled trial. BMC Public Health. 2019 Mar 1;19(1):255. doi: 10.1186/s12889-019-6574-y. PMID 30823909
- See also: short description in English — http://www.stopdia.fi/briefly-in-english